CLINICAL TRIAL: NCT02445248
Title: A Phase II, Single Arm, Multicenter Trial to Determine the Efficacy and Safety of CTL019 in Adult Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of Efficacy and Safety of CTL019 in Adult DLBCL Patients
Acronym: JULIET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019C2201; 2014-003060-20 (EudraCT Number)
Expanded Access: NCT03601442 (Available)
Record Dates: First submitted 2015-05-05; First posted 2015-05-15 (Estimated); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: Diffuse large B-cell lymphoma; DLBCL; Relapsed/refractory; CTL019; CART19; CART; CAR T cells; Chimeric antigen receptor
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (Experimental): Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel.
  Interventions: Biological: Tisagenlecleucel; Drug: Lymphodepleting chemotherapy

INTERVENTIONS:
Biological: Tisagenlecleucel — The target dose of CTL019 transduced cells for adult patients consisted of a single infusion of 5 x 10^8 viable CTL019 transduced cells, which was administered via intravenous infusion. The acceptable dose range was 1 - 5x10^8 viable CTL019 transduced cells.
  Other Names: CTL019
Drug: Lymphodepleting chemotherapy — Prior to CTL019 cell infusion, an additional lymphodepleting chemotherapy cycle was planned. The use of any additional bridging therapy prior to the recommended lymphodepleting chemotherapy was at the discretion of the investigator and dependent on the patient's disease burden. Lymphodepleting chemotherapy was started 14 to 5 days before CTL019 infusion (D1) to allow for at least 48 hours from last dose of lymphodepleting chemotherapy to CTL019 infusion. The lymphodepleting regimen was: Fludarabine (25 mg/m^2 intravenously [i.v.] daily for 3 doses) and cyclophosphamide (250 mg/m^2 i.v. daily for 3 doses starting with the first dose of fludarabine).

SUMMARY:
This is a multi-center, phase II study to determine the efficacy and safety of CTL019 in adult patients with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
This was a single arm, open-label, multi-center, Phase II study conducted to determine the efficacy and safety of tisagenlecleucel in adult patients with r/r DLBCL. The study consisted of the following sequential periods: Screening, Pre-Treatment, Treatment and Primary follow-up, Secondary follow-up, Survival follow-up.

Patients were enrolled in 2 cohorts to receive one tisagenlecleucel infusion as follows:

* Main Cohort (patients treated with tisagenlecleucel manufactured at the Novartis manufacturing facility in Morris Plains, US, referred to as "US manufacturing facility") and
* Cohort A (patients treated with tisagenlecleucel manufactured at the Fraunhofer Institut für Zelltherapie, Leipzig, Germany, referred to as "EU manufacturing facility").

The study enrolled adult patients ≥ 18 years with histologically confirmed relapsed or refractory (r/r) DLBCL after ≥ 2 lines of chemotherapy, with a life expectancy of ≥ 12 weeks and not eligible or not consenting to stem cell transplantation (SCT).

Patients had measurable disease at time of enrollment, adequate organ function and zero or one Eastern Cooperative Oncology Group performance status at screening. For each patient, the apheresis product of non-mobilized cells was received and accepted by the manufacturing site.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures
* Histologically confirmed DLBCL at last relapse(by central pathology review before enrolment.

  .- Relapsed or refractory disease after ≥2 lines of chemotherapy including rituximab and anthracycline and either having failed autologous Hematopoietic stem cell transplantation (ASCT), or being ineligible for or not consenting to ASCT
* Measurable disease at time of enrollment
* Life expectancy ≥12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening
* Adequate organ function:

  * Renal function defined as:

    * A serum creatinine of ≤1.5 x Upper Limit of Normal ULN OR
    * Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73 m^2
  * Liver function defined as:

    * Alanine Aminotransferase (ALT) ≤ 5 times the Upper Limit of Normal (ULN) for age
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
  * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air
  * Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA)
  * Adequate bone marrow reserve without transfusions defined as:

    * Absolute neutrophil count (ANC) > 1.000/mm^3
    * Absolute lymphocyte count (ALC) ≥ 300/mm^3 and absolute number of CD3+ T cells > 150/mm^3
    * Platelets ≥ 50.000//mm^3
    * Hemoglobin > 8.0 g/dl
  * Must have an apheresis product of non-mobilized cells accepted for manufacturing
  * Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) and all male participants must agree to use highly effective methods of contraception for at least 12 months following CTL019 infusion and until CAR T cells are no longer present by PCR on two consecutive tests

Exclusion Criteria:

* Prior treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy
* Treatment with any prior gene therapy product
* Active Central Nervous System (CNS) involvement by malignancy
* Prior allogeneic HSCT
* Eligible for and consenting to HSCT
* Chemotherapy other than lymphodepleting chemotherapy within 2 weeks of infusion
* Investigational medicinal product within the last 30 days prior to screening
* The following medications are excluded:

  * Steroids: Therapeutic doses of steroids must be stopped >72 hours prior to leukapheresis and >72 hours prior to CTL019 infusion. However, the following physiological replacement doses of steroids are allowed: < 12 mg/m^2/day hydrocortisone or equivalent
  * Immunosuppression: Any other immunosuppressive medication must be stopped ≥2 weeks prior to leukapheresis and ≥ 2 weeks prior to CTL019 infusion. This could include check point inhibitors (monoclonal antibodies and small molecule modulators)
  * Antiproliferative therapies other than lymphodepleting chemotherapy within two weeks of leukapheresis and 2 weeks prior to infusion
* Short acting drugs used to treat leukemia or lymphoma (e.g. tyrosine kinase inhibitors, and hydroxyurea) must be stopped > 72 hour prior to leukapheresis and > 72 hours prior to CTL019 infusion
* Other cytotoxic drugs, including low dose daily or weekly maintenance chemotherapy, must not be given within 2 weeks prior to leukapheresis and within 2 weeks prior to CTL019 infusion
* Fludarabine may be associated with prolonged lymphopenia. This should be taken into consideration when evaluating the optimal timing for leukapheresis collection.

  * Antibody use including anti-CD20 therapy within 4 weeks prior to infusion or 5 half-lives of the respected antibody, whichever is longer
  * CNS disease prophylaxis must be stopped > 1 week prior to CTL019 infusion (e.g. intrathecal methotrexate)
* Prior radiation therapy within 2 weeks of infusion
* Active replication of or prior infection with hepatitis B or active hepatitis C( HCV RNA positive )
* HIV positive patients
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 6 months prior to screening
* Previous or concurrent malignancy with the following exceptions:

  * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
  * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
  * A primary malignancy which has been completely resected and in complete remission for ≥ 5 years
* Pregnant or nursing (lactating) women. NOTE: female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 24 hours before lymphodepletion
* Intolerance to the excipients of the CTL019 cell product
* Cardiac arrhythmia not controlled with medical management
* Prior treatment with any adoptive T cell therapy
* Patients with T-cell rich/histiocyte rich large B-cell lymphoma (THRBCL), primary cutaneous large B-cell lymphoma, primary mediastinal B-cell lymphoma (PMBCL), EBV positive DLBCL of the elderly, Richter's transformation, and Burkitt lymphoma
* Patients with active neurological auto immune or inflammatory disorders (e.g. Guillain Barre Syndrome, Amyptrophic Lateral Sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- United States (12):
  - UCSF Medical Center ., San Francisco, California
  - Emory University School of Medicine/Winship Cancer Institute SC CTL019, Atlanta, Georgia
  - University of Chicago Medical Center Hematology and Oncology SC - CTL019B2207J, Chicago, Illinois
  - University of Kansas Cancer Center SC - CTL019C2201, Westwood, Kansas
  - Sidney Kimmel Comprehensive Cancer Center SC-2, Baltimore, Maryland
  - Uni of Michigan Health System SC CTL019, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medical College, New York, New York
  - The Ohio State University James Cancer Hospital &, Columbus, Ohio
  - Oregon Health Sciences University Oregon Health & Sci Uni, Portland, Oregon
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center SC, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Camperdown
- Novartis Investigative Site, Vienna, Austria
- Canada (2):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Pierre-Bénite, France
- Germany (2):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Milan, MI, Italy
- Japan (3):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Maziarz RT, Bishop MR, Tam CS, Borchmann P, Worel N, McGuirk JP, Holte H, Waller EK, Jaglowski S, Andreadis C, Foley SR, Westin JR, Fleury I, Ho PJ, Mielke S, Teshima T, Janakiram M, Hsu J, Izutsu K, Kersten MJ, Ghosh M, Wagner-Johnston N, Kato K, Corradini P, Ma W, Han X, Nuortti M, Awasthi R, Mundt KE, Majdan M, Maier HJ, Jegerlehner A, Salles G, Schuster SJ. Five-Year Analysis of the JULIET Trial of Tisagenlecleucel in Patients With Relapsed/Refractory Large B-Cell Lymphoma. J Clin Oncol. 2026 Jan 10;44(2):86-91. doi: 10.1200/JCO-25-00507. Epub 2025 Nov 18. PMID 41252666
- [Derived] Cartron G, Fox CP, Liu FF, Kostic A, Hasskarl J, Li D, Bonner A, Zhang Y, Maloney DG, Kuruvilla J. Matching-adjusted indirect treatment comparison of chimeric antigen receptor T-cell therapies for third-line or later treatment of relapsed or refractory large B-cell lymphoma: lisocabtagene maraleucel versus tisagenlecleucel. Exp Hematol Oncol. 2022 Mar 25;11(1):17. doi: 10.1186/s40164-022-00268-z. PMID 35337365
- [Derived] Frigault MJ, Dietrich J, Gallagher K, Roschewski M, Jordan JT, Forst D, Plotkin SR, Cook D, Casey KS, Lindell KA, Depinho GD, Katsis K, Elder EL, Leick MB, Choi B, Horick N, Preffer F, Saylor M, McAfee S, O'Donnell PV, Spitzer TR, Dey B, DeFilipp Z, El-Jawahri A, Batchelor TT, Maus MV, Chen YB. Safety and efficacy of tisagenlecleucel in primary CNS lymphoma: a phase 1/2 clinical trial. Blood. 2022 Apr 14;139(15):2306-2315. doi: 10.1182/blood.2021014738. PMID 35167655
- [Derived] Schuster SJ, Tam CS, Borchmann P, Worel N, McGuirk JP, Holte H, Waller EK, Jaglowski S, Bishop MR, Damon LE, Foley SR, Westin JR, Fleury I, Ho PJ, Mielke S, Teshima T, Janakiram M, Hsu JM, Izutsu K, Kersten MJ, Ghosh M, Wagner-Johnston N, Kato K, Corradini P, Martinez-Prieto M, Han X, Tiwari R, Salles G, Maziarz RT. Long-term clinical outcomes of tisagenlecleucel in patients with relapsed or refractory aggressive B-cell lymphomas (JULIET): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2021 Oct;22(10):1403-1415. doi: 10.1016/S1470-2045(21)00375-2. Epub 2021 Sep 10. PMID 34516954
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Westin JR, Kersten MJ, Salles G, Abramson JS, Schuster SJ, Locke FL, Andreadis C. Efficacy and safety of CD19-directed CAR-T cell therapies in patients with relapsed/refractory aggressive B-cell lymphomas: Observations from the JULIET, ZUMA-1, and TRANSCEND trials. Am J Hematol. 2021 Oct 1;96(10):1295-1312. doi: 10.1002/ajh.26301. Epub 2021 Aug 13. PMID 34310745
- [Derived] Schuster SJ, Maziarz RT, Rusch ES, Li J, Signorovitch JE, Romanov VV, Locke FL, Maloney DG. Grading and management of cytokine release syndrome in patients treated with tisagenlecleucel in the JULIET trial. Blood Adv. 2020 Apr 14;4(7):1432-1439. doi: 10.1182/bloodadvances.2019001304. PMID 32271899
- [Derived] Maziarz RT, Schuster SJ, Romanov VV, Rusch ES, Li J, Signorovitch JE, Maloney DG, Locke FL. Grading of neurological toxicity in patients treated with tisagenlecleucel in the JULIET trial. Blood Adv. 2020 Apr 14;4(7):1440-1447. doi: 10.1182/bloodadvances.2019001305. PMID 32271898
- [Derived] Maziarz RT, Waller EK, Jaeger U, Fleury I, McGuirk J, Holte H, Jaglowski S, Schuster SJ, Bishop MR, Westin JR, Mielke S, Teshima T, Bachanova V, Foley SR, Borchmann P, Salles GA, Zhang J, Tiwari R, Pacaud LB, Ma Q, Tam CS. Patient-reported long-term quality of life after tisagenlecleucel in relapsed/refractory diffuse large B-cell lymphoma. Blood Adv. 2020 Feb 25;4(4):629-637. doi: 10.1182/bloodadvances.2019001026. PMID 32074277
- [Derived] Awasthi R, Pacaud L, Waldron E, Tam CS, Jager U, Borchmann P, Jaglowski S, Foley SR, van Besien K, Wagner-Johnston ND, Kersten MJ, Schuster SJ, Salles G, Maziarz RT, Anak O, Del Corral C, Chu J, Gershgorin I, Pruteanu-Malinici I, Chakraborty A, Mueller KT, Waller EK. Tisagenlecleucel cellular kinetics, dose, and immunogenicity in relation to clinical factors in relapsed/refractory DLBCL. Blood Adv. 2020 Feb 11;4(3):560-572. doi: 10.1182/bloodadvances.2019000525. PMID 32045475
- [Derived] Bishop MR, Maziarz RT, Waller EK, Jager U, Westin JR, McGuirk JP, Fleury I, Holte H, Borchmann P, Del Corral C, Tiwari R, Anak O, Awasthi R, Pacaud L, Romanov VV, Schuster SJ. Tisagenlecleucel in relapsed/refractory diffuse large B-cell lymphoma patients without measurable disease at infusion. Blood Adv. 2019 Jul 23;3(14):2230-2236. doi: 10.1182/bloodadvances.2019000151. PMID 31332046
- [Derived] Schuster SJ, Bishop MR, Tam CS, Waller EK, Borchmann P, McGuirk JP, Jager U, Jaglowski S, Andreadis C, Westin JR, Fleury I, Bachanova V, Foley SR, Ho PJ, Mielke S, Magenau JM, Holte H, Pantano S, Pacaud LB, Awasthi R, Chu J, Anak O, Salles G, Maziarz RT; JULIET Investigators. Tisagenlecleucel in Adult Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2019 Jan 3;380(1):45-56. doi: 10.1056/NEJMoa1804980. Epub 2018 Dec 1. PMID 30501490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 participants were infused in this study: 99 in the Main Cohort and 16 in Cohort A.
Pre-assignment Details: After informed consent/assent was obtained, and prior to infusion, participants underwent a routine lymphodepleting therapy, 14 to 5 days before CTL019 infusion.
  There were 27 centers across 10 countries for this trial.
Groups:
- Tisagenlecleucel - Main Cohort: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Novartis manufacturing facility in Morris Plains, US.
- Tisagenlecleucel Cohort A: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Fraunhofer Institut für Zelltherapie, Leipzig, Germany.
Period: Overall Study
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel Cohort A
Started (Started = Infused) | 99 | 16
Completed (Completed = Study follow-up completed) | 26 | 3
Not Completed | 73 | 13
Not completed — Death | 45 | 12
Not completed — Progressive disease | 13 | 1
Not completed — Subject decision | 8 | 0
Not completed — Physician Decision | 5 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel Cohort A | Total
Number analyzed (Participants) | 99 | 16 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.09) | 51.1 (12.98) | 53.8 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 8 | 44
  Male | 63 | 8 | 71
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 83 | 15 | 98
  Asian | 10 | 0 | 10
  Black | 4 | 0 | 4
  Other | 2 | 1 | 3
ECOG performance status [Number; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance status is a numbering scale used in Oncology w to define the population of patients to study in the trial and guide physicians who enroll patients into those studies. The lower the number the better the performance status of the patient, where 0: Fully active, able to carry on all pre-disease performance without restriction. ECOG Performance status of 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG status of 0 | 54 | 11 | 65
    ECOG status of 1 | 45 | 5 | 50

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Independent Review Committee (IRC) in Main Cohort
Description: ORR, which includes complete response (CR) and partial response (PR) in the Main cohort as determined by IRC assessment. ORR is the percentage of participants with a best overall disease response of CR or PR, where the best overall disease response is defined as the best disease response recorded from CTL019 infusion until progressive disease or start of new anticancer therapy (including ASCT), whichever comes first.
  Response was assessed according to Evaluation Criteria in diffuse large B cell lymphoma studies (based on Cheson Response criteria and the Lugano Classification (2014))
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised of all patients in the Main cohort who received infusion of tisagenlecleucel.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tisagenlecleucel - Main Cohort
Number analyzed (Participants) | 99
Percentage of participants | 54.5 [44.2 to 64.6]

2. Secondary Outcome: Overall Response Rate (ORR) Per Independent Review Committee (IRC) in Cohort A & in All Patients
Description: ORR, which includes complete response (CR) and partial response (PR) in the Main cohort as determined by IRC assessment. ORR is the percentage of participants with a best overall disease response of CR or PR, where the best overall disease response is defined as the best disease response recorded from CTL019 infusion until progressive disease or start of new anticancer therapy (including ASCT), whichever comes first.
Time Frame: 5 years
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Tisagenlecleucel - Cohort A: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Fraunhofer Institut für Zelltherapie, Leipzig, Germany.
- Tisagenlecleucel - All Patients: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Novartis manufacturing facility in Morris Plains, US and at the Fraunhofer Institut für Zelltherapie, Leipzig, Germany.
Arm/Group | Tisagenlecleucel - Cohort A | Tisagenlecleucel - All Patients
Number analyzed (Participants) | 16 | 115
Percentage of participants | 43.8 [19.8 to 70.1] | 53.0 [43.5 to 62.4]

3. Secondary Outcome: Time to Response (TTR) as Assessed by Independent Review Committee (Main Cohort & All Patients)
Description: TTR is the time between date of CTL019 infusion until first documented response (CR or PR).
Time Frame: up to approx. 3.3 months
Population: Full Analysis Set (FAS): Comprised all patients in the Main cohort who received infusion of tisagenlecleucel.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel - All Patients
Number analyzed (Participants) | 99 | 115
Months | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.0]

4. Secondary Outcome: Duration of Overall Response (DOR) Per IRC
Description: DOR is the time from achievement of CR or PR, whichever occurs first, to relapse or death due to diffuse large B-cell lymphoma (DLBCL).
Time Frame: up to approx. 60.1 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel and who achieved a completer response (CR) or a partial response (PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel - Cohort A | Tisagenlecleucel - All Patients
Number analyzed (Participants) | 54 | 7 | 61
Months | NA [10.0 to NA] — NA: The Median and the upper limit of Confidence Interval could not be reached because fewer than half of the patients experienced an event | NA [1.2 to NA] — NA: The Median and the upper limit of Confidence Interval could not be reached because fewer than half of the patients experienced an event | NA [10.0 to NA] — NA: The Median and the upper limit of Confidence Interval could not be reached because fewer than half of the patients experienced an event

5. Secondary Outcome: Event Free Survival (EFS) Per Independent Review Committee
Description: EFS is the time from date of CTL019 infusion to the date of first documented disease progression or relapse, new treatment for lymphoma or death due to any cause.
Time Frame: up to approx. 61 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel - Cohort A | Tisagenlecleucel - All Patients
Number analyzed (Participants) | 99 | 16 | 115
Months | 2.8 [2.2 to 3.5] | 2.1 [1.0 to 3.1] | 2.8 [2.1 to 3.1]

6. Secondary Outcome: Progression Free Survival (PFS) Per Independent Review Committee
Description: PFS is the time from date of CTL019 infusion to the date of first documented disease progression or death due to any cause.
Time Frame: up to approx. 61 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Tisagenlecleucel - All Patients: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at a US facility and an EU facility (Fraunhofer Institut für Zelltherapie, Leipzig, Germany).
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel - Cohort A | Tisagenlecleucel - All Patients
Number analyzed (Participants) | 99 | 16 | 115
Months | 3.0 [2.4 to 6.2] | 2.9 [1.0 to NA] — NA: The upper limit of the Confidence Interval could ne be reached because there were not enough events to estimate the time to the later events. | 2.9 [2.3 to 5.2]

7. Secondary Outcome: Overall Survival (OS) Per Independent Review Committee
Description: OS is the time from date of CTL019 infusion to the date of death due to any cause.
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tisagenlecleucel - Main Cohort | Tisagenlecleucel - Cohort A | Tisagenlecleucel - All Patients
Number analyzed (Participants) | 99 | 16 | 115
Months | 12.5 [7.2 to 34.2] | 5.9 [3.1 to 19.2] | 11.1 [6.6 to 23.9]

8. Secondary Outcome: Pharmacokinetics (Pk): Cmax
Description: Cmax is the maximum (peak) observed in peripheral blood or other body fluid drug concentration after single dose administration. Cmax, based on the transgene level data by qPCR, was summarized by Month 3 response, per Independent Review Committee assessment. The reported Cmax is the summary of maximum level observed based on the data from each patient and based on all the data that's been collected for up to 60 months in a patient.
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel with valid PK assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug
Groups:
- Tisagenlecleucel - Main Cohort: CR/PR; Tisagenlecleucel - Main Cohort: SD/PD/UNK: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Novartis manufacturing facility in Morris Plains, US.
- Tisagenlecleucel - Cohort A: CR/PR; Tisagenlecleucel - Cohort A: SD/PD/UNK: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Fraunhofer Institut für Zelltherapie, Leipzig, Germany.
Arm/Group | Tisagenlecleucel - Main Cohort: CR/PR | Tisagenlecleucel - Main Cohort: SD/PD/UNK | Tisagenlecleucel - Cohort A: CR/PR | Tisagenlecleucel - Cohort A: SD/PD/UNK
Number analyzed (Participants) | 40 | 56 | 4 | 11
copies/ug | 5570 (271.3) | 4690 (481.1) | 14300 (67.5) | 6950 (109.3)

9. Secondary Outcome: Pharmacokinetics (Pk): Tmax
Description: Tmax is the time to reach maximum (peak) peripheral blood or other body fluid drug concentration after single dose administration (days). Tmax, based on the transgene level data by qPCR, was summarized by Month 3 response, per Independent Review Committee assessment. The time frame of 60 months refers to the duration for which the data were reviewed to identify the time of Cmax for this measure.
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel with valid PK assessments.
Measure: Median (Full Range); unit: days
Arm/Group | Tisagenlecleucel - Main Cohort: CR/PR | Tisagenlecleucel - Main Cohort: SD/PD/UNK | Tisagenlecleucel - Cohort A: CR/PR | Tisagenlecleucel - Cohort A: SD/PD/UNK
Number analyzed (Participants) | 40 | 56 | 4 | 11
days | 9.84 [5.78 to 27.7] | 8.95 [0.994 to 26.7] | 6.95 [5.94 to 8.96] | 6.93 [6.67 to 10.9]

10. Secondary Outcome: Pharmacokinetics (Pk): AUC0-28d and AUC0-84d
Description: The AUC from time zero to day 28 and 84 or other disease assessment days, in peripheral blood. AUC0-28d and AUC0-84d, based on the transgene level data by qPCR, were summarized by Month 3 response, per Independent Review Committee assessment.
Time Frame: 0 - 28 days after infusion for AUC0-28d, 0 - 84 days after infusion for AUC0-84d
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel with valid PK assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug*days
Groups:
- Tisagenlecleucel - CR/PR; Tisagenlecleucel - Main Cohort: SD/PD/UNK: Adult patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who received tisagenlecleucel manufactured at the Novartis manufacturing facility in Morris Plains, US.
Arm/Group | Tisagenlecleucel - CR/PR | Tisagenlecleucel - Main Cohort: SD/PD/UNK | Tisagenlecleucel - Cohort A: CR/PR | Tisagenlecleucel - Cohort A: SD/PD/UNK
Number analyzed (Participants) | 40 | 59 | 4 | 12
copies/ug*days
  AUC0-28d: number analyzed (Participants) | 39 | 50 | 4 | 12
  AUC0-28d | 58000 (182.1) | 49900 (388.5) | 141000 (78.2) | 63700 (134.2)
  AUC0-84d: number analyzed (Participants) | 39 | 24 | 4 | 5
  AUC0-84d | 102000 (171.7) | 92900 (165.4) | 206000 (76.7) | 142000 (61.3)

11. Secondary Outcome: Pharmacokinetics (Pk): T1/2
Description: T1/2 is the half-life associated with the disposition phase slopes (alpha, beta, gamma etc.) of a semi logarithmic concentration-time curve in peripheral blood. T1/2, based on the transgene level data by qPCR, was summarized by Month 3 response, per Independent Review Committee assessment. This time frame of 60 months reflects the maximum duration up to which the transgene levels were collected to measure the half life.
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel with valid PK assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Tisagenlecleucel - Main Cohort: CR/PR | Tisagenlecleucel - Main Cohort: SD/PD/UNK | Tisagenlecleucel - Cohort A: CR/PR | Tisagenlecleucel - Cohort A: SD/PD/UNK
Number analyzed (Participants) | 28 | 40 | 3 | 9
days | 167 (355.3) | 10.9 (205.4) | 59.4 (30402.1) | 15.6 (163.5)

12. Secondary Outcome: Pharmacokinetics (Pk): Clast
Description: Clast is the last observed quantifiable concentration in peripheral blood. Clast, based on the transgene level data by qPCR, was summarized by Month 3 response, per Independent Review Committee assessment. This time frame reflects maximum duration of 60 months up to which the transgene levels were collected.
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel with valid PK assessments.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | Tisagenlecleucel - Main Cohort: CR/PR | Tisagenlecleucel - Main Cohort: SD/PD/UNK | Tisagenlecleucel - Cohort A: CR/PR | Tisagenlecleucel - Cohort A: SD/PD/UNK
Number analyzed (Participants) | 40 | 55 | 4 | 12
copies/ug | 181 (114.4) | 332 (430.9) | 272 (30.6) | 386 (540.9)

13. Secondary Outcome: Pharmacokinetics (Pk): Tlast
Description: Tlast is the time of last observed quantifiable concentration in peripheral blood. Tlast, based on the transgene level data by qPCR, was summarized by Month 3 response, per Independent Review Committee assessment. This time frame reflects maximum duration of 60 months up to which the transgene levels were collected.
Time Frame: 60 months
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel with valid PK assessments.
Measure: Median (Full Range); unit: days
Arm/Group | Tisagenlecleucel - Main Cohort: CR/PR | Tisagenlecleucel - Main Cohort: SD/PD/UNK | Tisagenlecleucel - Cohort A: CR/PR | Tisagenlecleucel - Cohort A: SD/PD/UNK
Number analyzed (Participants) | 40 | 55 | 4 | 12
days | 930 [18.0 to 1830] | 41.9 [0.994 to 1480] | 1040 [17.1 to 1830] | 59.4 [26.8 to 126]

14. Secondary Outcome: Incidence of Immunogenicity to CTL019
Description: This is defined as the percentage of participants who tested positive for anti-mCAR19 antibodies at any time post-baseline, reported by complete response (CR), partial response (PR), Stable disease (SD), progressive disease (SD), Unknown for all participants who received with tisagenlecleucel.
Time Frame: pre-infusion and at any time point post-baseline, up to duration of the study, up to 5 years
Population: Full Analysis Set (FAS): Comprised all patients who received infusion of tisagenlecleucel.
Measure: Count of Participants; unit: Participants
Groups:
- Tisagenlecleucel - All Participants Response: Participants with complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) and unknown (UNK) response post-tisagenlecleucel infusion.
Arm/Group | Tisagenlecleucel - All Participants Response
Number analyzed (Participants) | 115
Participants
  Complete response: number analyzed (Participants) | 37
  Complete response | 36
  Partial response: number analyzed (Participants) | 7
  Partial response | 6
  Stable disease: number analyzed (Participants) | 1
  Stable disease | 1
  Progressive disease: number analyzed (Participants) | 54
  Progressive disease | 50
  Unknown: number analyzed (Participants) | 16
  Unknown | 14
  All Participants | 107

15. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths, which include post-treatment survival follow-up deaths, were collected during the post-infusion period (starting at the day of first infusion) until the end of the study, approx. 61 months.
  All deaths refers to the sum of on-treatment deaths and post-treatment survival follow-up deaths up to approx. 61 months.
Time Frame: On-treatment deaths: Up to 61 months; Post-treatment survival follow-up deaths: Up to approx. 61 months
Population: Clinical Database Population: all infused participants in the Study.
Measure: Number; unit: Participants
Arm/Group | Tisagenlecleucel - Main Cohort
Number analyzed (Participants) | 115
Participants
  On-treatment deaths include post-treatment survival follow-up deaths | 76
  All deaths | 76

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected during the post-infusion period (starting at the day of 1st infusion until the end of the study), up to maximum duration of 61 months for each patient. Deaths were collected at all points post-infusion until the patient completed the study duration (60 months) or further safety follow-up under the study protocol. Therefore on-treatment deaths include post-infusion deaths until Last patient Last Visit (LPLV).
Description: AE is any sign or symptom that occurs during the post-infusion period (starting at the day of first infusion of CTL019 until the end of the study) and safety follow-up. Deaths in post treatment survival follow-up are not considered Adverse Events while still included in the All-Cause Mortality table. Adverse
  Adverse event data were pre-specified in the secondary objectives to be analyzed for all treated patients as one group.
Arm/Group | Tisagenlecleucel - All Patients
All-Cause Mortality (participants affected / at risk) | 76/115
Serious Adverse Events (participants affected / at risk) | 84/115
Other Adverse Events (participants affected / at risk) | 113/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel - All Patients (N=115)
Bone marrow failure (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 4
Influenza like illness (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 3
Pyrexia (General disorders) | 9
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 31
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cerebral toxoplasmosis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 3
Corynebacterium infection (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 9
Pneumonia aspiration (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Systemic infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Refractory cytopenia with multilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute polyneuropathy (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 4
Ischaemic cerebral infarction (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel - All Patients (N=115)
Anaemia (Blood and lymphatic system disorders) | 55
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Tachycardia (Cardiac disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 36
Dry mouth (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 33
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 8
Chills (General disorders) | 14
Fatigue (General disorders) | 28
Influenza like illness (General disorders) | 9
Oedema peripheral (General disorders) | 17
Pain (General disorders) | 6
Pyrexia (General disorders) | 35
Cytokine release syndrome (Immune system disorders) | 47
Hypogammaglobulinaemia (Immune system disorders) | 10
Influenza (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 9
Pneumonia (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 15
Urinary tract infection (Infections and infestations) | 10
Blood creatinine increased (Investigations) | 12
Blood immunoglobulin G decreased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 40
Platelet count decreased (Investigations) | 38
Weight decreased (Investigations) | 14
White blood cell count decreased (Investigations) | 41
Decreased appetite (Metabolism and nutrition disorders) | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 19
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 24
Anxiety (Psychiatric disorders) | 11
Confusional state (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT02445248/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT02445248/SAP_001.pdf